CLINICAL TRIAL: NCT00327639
Title: Factors Promoting Increased Rate and Success of Pregnancy in the Thalassemia Population in Toronto
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Other Study IDs: 00000
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2006-05-18 (Estimated); Status verified 2005-07

CONDITIONS: Thalassemia; Fertility; Pregnancy
MeSH Terms: conditions — Thalassemia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Treatment of patients with beta thalassemia in North America has altered dramatically during the past 40 years, with improvements in transfusion therapy and introduction of iron chelation therapy. Thalassemia patients now enjoy an increased life expectancy to the fifth and sixth decades of life, with fertility and childbearing becoming important issues. Data regarding this important topic remain limited, without clear data regarding iron control including serial assessment of hepatic iron concentration, the need for assistance in becoming pregnant, and use of iron chelating agents during pregnancy. As the life expectancy increases and overall health improves in thalassemia, clear data on fertility, pregnancy complications, and the effect of pregnancy on maternal health in thalassemia patients are necessary since these will have a direct impact on patient care, quality of life, and patient expectations.

ELIGIBILITY:
Inclusion Criteria:

* Thalassemia, thalassemia intermedia or E-thalassemia patients in Toronto
* Subject has attempted conception

Exclusion Criteria:

* Subject has any other form of blood disease
* Subject has not attempted conception

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2005-07

CONTACTS AND LOCATIONS:
Overall Officials: Nancy F Olivieri, MD, Principal Investigator — University Health Network, Toronto General Hospital
Locations (1):
- University Health Network, Toronto General Hospital, Toronto, Ontario, Canada